CLINICAL TRIAL: NCT01697150
Title: Systems Approach to Closed-Loop Control of Type 1 Diabetes at Home
Brief Title: Outpatient Control-to-Range: System and Monitoring Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: University of California, Santa Barbara (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Jordan Pinsker, Director of Clinical Research and Diabetes Technology, Sansum Diabetes Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDRF 22-2011-649 SB
Record Dates: First submitted 2012-04-19; First posted 2012-10-02 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; closed loop artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control to Range Testing (Experimental): Subjects will spend two nights in a non hospital setting while the DiAs Diabetes Assistant Wearable Artificial Pancreas Platform is remotely monitored from an adjacent room. DiAs Diabetes Assistant Wearable Artificial Pancreas Platform is composed of an Android-based cell phone platform operating with a DexCom sensor, OmniPod Insulin Management System and an Insulet iDex remote controller. Communication runs on a tablet. The Control to Range software will be capable of transmitting patient state data to a remote monitoring device. The subject will be trained on the open loop features of the cell phone platform user interface: DexCom displays, Insulin injection history display, bolus function. The subject may use the study pump per his/her usual home regimen and may make adjustments to his/her insulin based on symptoms or SMBG readings.
  Interventions: Device: DiAs Diabetes Assistant Wearable Artificial Pancreas Platform

INTERVENTIONS:
Device: DiAs Diabetes Assistant Wearable Artificial Pancreas Platform — Subjects will spend two nights in a non hospital setting while the Artificial Pancreas Device System is remotely monitored from an adjacent room. Artificial Pancreas Device System is composed of an Android-based cell phone platform operating with a DexCom sensor, OmniPod Insulin Management System and an Insulet iDex remote controller. Communication runs on a tablet. The Control to Range software will be capable of transmitting patient state data to a remote monitoring device. The subject will be trained on the open loop features of the cell phone platform user interface: DexCom displays, Insulin injection history display, bolus function. The subject may use the study pump per his/her usual home regimen and may make adjustments to his/her insulin based on symptoms or SMBG readings.

SUMMARY:
Automated closed-loop control (CLC) of blood glucose, known as "artificial pancreas" (AP) can have tremendous impact on the health and lives of people with type 1 diabetes (T1DM). The investigators inter-institutional and international research team has been on the forefront of CLC developments since the beginning of the JDRF Artificial Pancreas initiative in 2006. Thus far, the investigators have conducted three closed-loop control clinical trials (totaling 60 subjects with T1DM), which demonstrated significantly more time in an acceptable "target" blood glucose range during CLC, and significantly fewer hypoglycemic events during CLC compared to open loop. The investigators overall objective is to sequentially test, validate, obtain regulatory approval for, and deploy at home, a closed-loop Control-to-Range (CTR) system comprised of two algorithmic components: a Safety Supervision Module (SSM) and a Hypoglycemia Mitigation Module (HMM). The SSM will monitor the safety of the subject's continuous subcutaneous insulin infusion pump (CSII) to prevent hypoglycemia and will also monitor the integrity of continuous glucose monitor (CGM) data for signal sensor deviations or loss of sensitivity. The HMM will be responsible for the optimal regulation of postprandial hyperglycemic excursions through correction boluses.

This study will test the ability of AP Platform to (1) run CTR in an outpatient setting, and (2) be remotely monitored. Specifically, this study involves studying adults with T1DM who are experienced insulin pump users. Subjects will spend two nights (-42 hours) in a local hotel, during which the AP Platform will be remotely monitored in an adjacent hotel room for validation that remote system monitoring can successfully occur. During the study, study subject will be responsible for. operating the CTR system with nursing and technicians available

DETAILED DESCRIPTION:
I.A. PURPOSE/OBJECTIVES

1. Primary objective The purpose of this pilot study is to test a closed-loop Control-to-Range (CTR) system in a semi-controlled environment and especially to evaluate if the system can accurately collect data coming from patient inputs, insulin pump, and continuous glucose monitoring (CGM) device with more than 80% of time of use.
2. Secondary objectives

This pilot study will use a Artificial Pancreas Platform (AP Platform) cell phone/phone-based system to test an outpatient controller and remote monitoring as follows:

* test that the CTR system can be remotely monitored by nurses/physicians/ technicians to confirm appropriate functioning outside of the hospital setting
* test that the CTR system can be deployed, with appropriate subject response, outside of the hospital setting

I.B. STUDY DESIGN

This study is an early feasibility pilot trial with the principal goal is to validate an initial outpatient ready CTR system and its remote-monitoring capability. Therefore, this is an unblinded pilot study and no control group will be used.

ELIGIBILITY:
Inclusion Criteria:

1. ≥21 and <65 years old
2. Clinical diagnosis of type 1 diabetes mellitus:

   Criteria for documented hyperglycemia (at least 1 criterion must be met):
   * Fasting glucose ≥126 mg/dL - confirmed
   * Two-hour OGTT glucose ≥200 mg/dL - confirmed
   * HbA1c ≥6.5% documented by history - confirmed
   * Random glucose ≥200 mg/dL with symptoms
   * No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes

   Criteria for requiring insulin at diagnosis (at least 1 criterion must be met):
   * Participant required insulin at diagnosis and continually thereafter
   * Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
   * Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
3. Use of an insulin pump to treat his/her diabetes for at least 1 year
4. Actively using an insulin pump with bolus calculator feature including predefined parameters for carbohydrate ratio, insulin sensitivity factor, target BG and active insulin.
5. HbA1c between 6.0% - 9.0% as measured with DCA2000 or equivalent device
6. Not currently known to be pregnant, breast feeding, or intending to become pregnant (females)
7. Demonstration of proper mental status and cognition for the study
8. Willingness to avoid consumption of acetaminophen-containing products during the study interventions involving DexCom use
9. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study

Exclusion Criteria:

1. ≥21 and <65 years old
2. Clinical diagnosis of type 1 diabetes mellitus:

   * Criteria for documented hyperglycemia (at least 1 criterion must be met):

     * Fasting glucose ≥126 mg/dL - confirmed
     * Two-hour OGTT glucose ≥200 mg/dL - confirmed
     * HbA1c ≥6.5% documented by history - confirmed
     * Random glucose ≥200 mg/dL with symptoms
     * No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes
   * Criteria for requiring insulin at diagnosis (at least 1 criterion must be met):

     * Participant required insulin at diagnosis and continually thereafter
     * Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
     * Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
3. Use of an insulin pump to treat his/her diabetes for at least 1 year
4. Actively using an insulin pump with bolus calculator feature including predefined parameters for carbohydrate ratio, insulin sensitivity factor, target BG and active insulin.
5. HbA1c between 6.0% - 9.0% as measured with DCA2000 or equivalent device
6. Not currently known to be pregnant, breast feeding, or intending to become pregnant (females)
7. Demonstration of proper mental status and cognition for the study
8. Willingness to avoid consumption of acetaminophen-containing products during the study interventions involving DexCom use
9. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percent time of active CTR | 42 hours
  The main endpoint will be the percent time with all expected data from CGM, pump and patient manual inputs that should be available on Artificial Pancreas platform and monitoring stations. To be considered as successful, this percent time will have to reach more than 80% of total time of investigation.

SECONDARY OUTCOMES:
Frequency analysis of failed data caused by system components | 42 hours
  The failed data records will be compared to failure/missing data records from our past in-clinic studies
Frequency of inaccurate data caused by system components | 42 hours
  Continuous glucose sensor data will be compared with Hemocue data for accuracy.
Frequency analysis of lost data caused by system components | 42 hours
  The failure/missing data records will be compared to missing data records from our past in-clinic studies

CONTACTS AND LOCATIONS:
Overall Officials: Howard Zisser, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

REFERENCES:
- See also: http://www.sansum.org/research-trials/current-trials/ — http://www.sansum.org